CLINICAL TRIAL: NCT04718324
Title: Electronic Patient Reported Outcome Measures (ePROMs) in Patients With Breast Disease: An Open-label, Randomized Controlled Trial on Patient Reported Experience Measures (PREMs) and Effectivity (PREMs_PROMs)
Brief Title: PREMs on PROMs in Breast Disease (PREMs_PROMs)
Acronym: PREMs_PROMs
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Principal Investigator, Andreas Karakatsanis, Principal Investigator, Uppsala University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UUBreast02
Record Dates: First submitted 2020-12-26; First posted 2021-01-22 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Breast Disease; Breast Cancer; Breast Neoplasms
Keywords: Randomized Controlled Trial; PROMS; PREMS
MeSH Terms: conditions — Breast Diseases; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- e-PROMS (Experimental): Patients allocated to the e-PROMS arm will fill an online version of PROMS and then respond to the e-PREMS questionnaire.
  Interventions: Other: e-PROMS
- p-PROMS (Active Comparator): Patients allocated to the p-PROMS arm will fill in PROMS in paper form (p-PROMS) and then respond to the p-PREMS questionnaire.
  Interventions: Other: p-PROMS

INTERVENTIONS:
Other: e-PROMS — Participants randomised to the e-PROMS arm will receive a safe link to the e-PROMS and a unique identification number in the electronic form, so as to preserve anonymity. This is a one-time intervention
  Arms: e-PROMS
Other: p-PROMS — Participants randomised to the p-PROMS arm will receive the PROMS and PREMS questionnaires and a unique identification number in paper form.
  Arms: p-PROMS

SUMMARY:
In recent years, large interest in the conduct and focus of clinical trials has focused to patient related outcomes and value-based healthcare. Patient Reported Outcome MeasureS, (PROMs) has become one of the standard instruments used for measuring outcomes; multiple PROMS have been extensively validated and are used in many clinical studies, but also in clinical routine. Additionally, Patient Reported Experience MeasureS (PREMS) allow for real-time feedback on the integration of care and can subsequently drive changes in health provision systems. In the present trial, the mode of delivery of PROMS is examined in terms of effectivity and patient experience (PREMS) in the setting of breast disease.

DETAILED DESCRIPTION:
In recent years, large interest in the conduct and focus of clinical trials has focused to patient related outcomes and value-based healthcare. Patient Reported Outcome MeasureS, (PROMs) has become one of the standard instruments used for measuring outcomes; multiple PROMS have been extensively validated and are used in many clinical studies, but also in clinical routine. This is certainly the case for patients with breast disease, and in particular, breast cancer, where therapeutic advances in systemic and locoregional treatment have dramatically improved survival outcomes and shifted the interest in patient wellness, quality of life and health economy. However, their introduction and implementation require the development of certain logistics involving delivery to the patients, data procession and finally inclusion in patient journals and/or trial case report forms (CRFs).Additionally, Patient Reported Experience MeasureS (PREMS) allow for real-time feedback on the integration of care and can subsequently drive changes in health provision systems.

Currently, the paper-version of these PROMs, pPROMs, has been the standard version. With this comes some advantages, such as the ability to save and store filled PROMS, and for patients to fill them out when it suits them best, not having to answer all questions at once. At the same time, there are also disadvantages, such as that storing and processing the data is a tedious and resource-consuming task. Additionally, patients occasionally find it inconvenient to return the pPROMS by post; finally, the consumption of paper is not viewed as a environmentally friendly behaviour. At the same time and in the new era of digitalization, internet-based studies, such as surveys, become more popular. Most validated PROMS have been utilised in several occasions, and there is an effort for their standardisation in health care. These e-PROMs (electronic PROMs) seem to be more time-efficient since they do not have to be processed manually, but instead can be directly connected to digital systems which transform raw data (patient response) to big data and scores. It is also a more environment-friendly option since there is no need to print the questionnaires on paper or send them via mail to the patients and then back to the research centre. The question is how patients feel about these electronic versions and if their implementation may simplify PROMS, both for patients and healthcare givers and researchers alike. Even though the older generation at greater length is connected to the internet than before, and are more used to handling it, there are still those who are not comfortable with these new digital services.

Despite this being a reasonable hypothesis, no trials have examined this subject, that is to map the patients' attitudes toward participating in studies, nor which form is the preferred one, ePROMs or pPROMS. It would be reasonable to hypothesize that a more convenient mode of delivery would facilitate patients and would therefore increase response rates. Additionally, there is no randomized data on the optimal mode of PROMS delivery and process as far as monetary, personnel and structural resources are concerned

Reference population for the trial are women from the breast radiology unit, breast outpatient clinic and breast cancer patients from the oncology department of the participating sites. Patients will be asked to participate to this study through a letter sent they receive when receiving their appointment to the respective clinic/department. All patients are asked, regardless of diagnosis, sex or age; at this point, the researchers are not aware of individual information. If they consent, participants are randomised to either e-PROMs or pPROMs.

Trial hypothesis is that ePROMs are more convenient and time-efficient and that with these investigators can increase the response rate from 65% (which was observed in a pilot study previously conducted at the breast outpatient clinic at Uppsala University Hospital) to 80%.The trial is designed as a superiority trial to detect for a 0.15 difference between arms, with a 2-sided p-value=0.05 and 80% power. Sample size calculation was performed with (SampleSize4ClinicalTrials and TrialSize packages). This responds to 109 patients per arm. Patient allocation (1:1) is performed through permuted block randomisation performed on the R statistical software (randomizeR package) in blocks of 8.

Patients that provide oral and written consent for the trial are anonymised and receive a unique study number. They willingly provide contact details (address and e-mail address), in order to receive PROMS after randomization. Patients may decline mode of PROMS delivery, if they prefer otherwise. Patient preference is registered. In analyses, the "intention-to-treat" principle will be followed, but per protocol analyses is intended if the crossover is deemed significant (>10%).

Data process and analysis

Once filled out, the anonymised ePROMs will be automatically stored to the Uppsala University servers. They are extractable as a Microsoft Excel data sheet. pPROMS will be stored in paper form in a safe location at the participating site. All raw data from both arms will be transferred in an Excel database. This raw data will be processed through algorithms specific to each PROMS to allow for the calculation of the respective PROMS scores.

The time required for this procedure will be registered for statistical analyses.

Patient data to be utilised in the analysis is age and site of recruitment. Other data to be registered are monetary costs for pPROMS postal, monetary costs for pPROMS related consumable materials and hourly cost for the documentation and registration of PROMS in patient electronic journals.

Data and patient safety

Patient data will be treated according to the General Data Protection Regulation (GDPR). The trial is not expected to affect treatment of patients or affect diagnostic work-up or treatment modality. Participants will not receive monetary compensation. For participants that are wishing it, PROMS scores will be included in their journals.

Publication

Trial results are expected to be submitted for publication in peer-reviewed journals. Positive and negative results as well as subgroup analyses for primary characteristics such as patient age are expected to be reported.

ELIGIBILITY:
Inclusion Criteria:

* Patients seeking or being treated for perceived or verified, benign or malignant breast disease.
* Women undergoing screening mammography.

Exclusion Criteria:

* Linguistic barriers.
* Deprivation of liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Response rate | Up to 8 weeks after receiving the questionnaires
  Number of participants who answered the questionnaires divided by number of participants who were allocated to the respective arm. Analyses will be performed without and with "reminders", per intention-to-treat and per protocol.
Patient Reported Experience outcomes (PREMS) | Up to 8 weeks after receiving the questionnaires
  PREMS score per respective arm. The PREMS score will be standard Likert items ranging from 1 to 7 and 1 to 5, with higher scores meaning a better outcome. Analyses will be performed without and with "reminders", per intention-to-treat and per protocol.

SECONDARY OUTCOMES:
Time of response | Up to 8 weeks after receiving the questionnaires
  Average time of response per arm. Analyses will be performed without and with "reminders", per intention-to-treat and per protocol.
Procedure-related costs | Up to 8 weeks after receiving the questionnaires
  Monetary costs per arm, including direct monetary costs and working hours for researchers and healthcare professionals to obtain PROMS. Analyses will be performed without and with "reminders", per intention-to-treat and per protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Karakatsanis, PhD, Principal Investigator — Uppsala University Hospital
Locations (1):
- Uppsala University Hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 2 years after publication

REFERENCES:
- [Derived] Pantiora E, Hedman LC, Aristokleous I, Sjokvist O, Karakatsanis A, Schiza A. Effect of mode of delivery of patient reported outcomes in patients with breast disease: a randomised controlled trial. Int J Surg. 2024 Jan 1;110(1):176-182. doi: 10.1097/JS9.0000000000000815. PMID 37800546